CLINICAL TRIAL: NCT04871412
Title: Pioneering Pre- and Post-Operative Integrative Care to Improve Thoracic Cancer Quality of Care - The Thoracic Peri-Operative Integrative Surgical Care Evaluation (POISE) Trial - Stage III
Brief Title: The Thoracic Peri-Operative Integrative Surgical Care Evaluation Trial - Stage III
Acronym: POISE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: The Canadian College of Naturopathic Medicine (Other); Lotte & John Hecht Memorial Foundation (Other); The Centre for Health Innovation (Unknown); University of Ottawa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20200796-01H
Record Dates: First submitted 2021-04-12; First posted 2021-05-04 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer; Gastric Cancer; Esophageal Cancer
Keywords: Natural Health Products; Thoracic Cancer; Surgery; Integrative Care; Nutrition; Physical Activity; Psychological Health
MeSH Terms: conditions — Lung Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Motor Activity; Psychological Well-Being | interventions — Vitamin D; Fish Oils; Probiotics; Curcumin; Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrative Care (Treatment) (Experimental): Participants in the Integrative arm will receive standard surgical and oncologic care at The Ottawa Hospital plus complementary care guided by a naturopathic doctor at The Centre for Health Innovation
  Interventions: Dietary Supplement: Vitamin D3 Drops; Dietary Supplement: Coriolus Versicolor; Dietary Supplement: Trident SAP 66:33 Lemon; Dietary Supplement: Probiotic Pro12; Dietary Supplement: Provitalix Pure Whey Protein; Dietary Supplement: Theracurmin 2X; Dietary Supplement: Green Tea Extract; Other: Nutrition Recommendations; Other: Physical Activity Recommendations; Behavioral: Psychological Recommendations
- Standard Care (Control) (No Intervention): Participants in the control arm will receive standard surgical and oncologic care at The Ottawa Hospital

INTERVENTIONS:
Dietary Supplement: Vitamin D3 Drops — 1,000 - 10,000 units daily based on serum levels for the duration of the study
  Other Names: Vitamin D
  Arms: Integrative Care (Treatment)
Dietary Supplement: Coriolus Versicolor — 1.5g twice daily for the duration of the study
  Arms: Integrative Care (Treatment)
Dietary Supplement: Trident SAP 66:33 Lemon — 3g once daily for the duration of the study
  Other Names: Fish Oil
  Arms: Integrative Care (Treatment)
Dietary Supplement: Probiotic Pro12 — 12 billion colony forming units daily during the peri-operative period (approximately 1 month pre and post-surgery)
  Other Names: Probiotics
  Arms: Integrative Care (Treatment)
Dietary Supplement: Provitalix Pure Whey Protein — 1 scoop (22g) once daily during the peri-operative period (approximately 1 month pre and post-surgery) and during any adjuvant chemotherapy and radiation treatments
  Other Names: Protein Powder
  Arms: Integrative Care (Treatment)
Dietary Supplement: Theracurmin 2X — 1.2g twice daily after the peri-operative period. including during adjuvant chemotherapy and radiation
  Other Names: Curcumin
  Arms: Integrative Care (Treatment)
Dietary Supplement: Green Tea Extract — 700 mg twice daily after the peri-operative period. Will not be given during adjuvant radiation or chemotherapy treatments.
  Other Names: EGCG
  Arms: Integrative Care (Treatment)
Other: Nutrition Recommendations — Based on the Mediterranean diet and lower glycemic index foods
  Arms: Integrative Care (Treatment)
Other: Physical Activity Recommendations — 150 minutes moderate intensity aerobic exercise per week plus the addition of a resistance exercise program on 2 of those days
  Arms: Integrative Care (Treatment)
Behavioral: Psychological Recommendations — Activities with the intention of actively improving the participant's mental and emotional health
  Arms: Integrative Care (Treatment)

SUMMARY:
Despite enormous advances in thoracic surgery and oncology, two critical issues concern patients undergoing curative-intent surgery for lung, gastric and esophageal cancer: first, a majority (~60%) of patients experience minor and major adverse events occurring during and in the days following surgery; second, patients worry about the significant risk of cancer recurrence and mortality months to years after surgery. These issues, combined with side effects of chemotherapy and radiation, have detrimental effects on health-related quality of life (HRQoL). On a deeper level, there is the problem of an ongoing failure to integrate and evaluate the best of what complementary medicine has to offer surgical oncology care. Too many clinical trials focus on single agent therapies, rather than broad multi-faceted individualized and integrative care interventions that are used in real world settings.

The Thoracic POISE project has the overarching goal of improving care for thoracic cancer patients by impacting HRQoL, reducing surgical adverse events, prolonging overall survival and pioneering integrative care delivery.

ELIGIBILITY:
Inclusion criteria

• Adults eligible for complete resection of lung, gastric or esophageal cancer

Exclusion criteria

* Small cell, carcinoid, or gastrointestinal stromal (GIST) tumours
* Any wedge resections of lung cancer
* History of cancer with active treatment in the last 3 years (not including superficial bladder cancer or non-melanoma skin cancer)
* Patients currently receiving care guided by an ND or who have previously seen an ND in the last 3 months
* Pregnant or breastfeeding women*
* Any reason which, in the opinion of the Principal Investigator (or delegate), would prevent the subject from participating in the study
* Use of an investigational drug or participation in an investigational study within 30 days prior to starting the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Participant Recruitment Rates | At the end of recruitment (estimated 1 year)
  Measured by the number of people who are enrolled in the study compared to the total number screened.
Participant Retention Rates | 2 Years
  Measured by the number of people who enrol in the study but subsequently withdraw. These numbers will be compared between arms.
Cross-over and contamination in the control arm - Supplement usage | 1 Year
  Measured by the number of participants in the control arm who use the integrative interventions outlined in the protocol independent of a naturopathic doctor. Information on the number of supplements used and the length of use use will be collected at each standard of care visit.
Cross-over and contamination in the control arm - Mediterranean Diet Scores | 1 year
  Measured by the number of participants in the control arm who use the integrative interventions outlined in the protocol independent of a naturopathic doctor. Mediterranean diet scores (scale of 0-9) will be calculated in the control group using the Harvard Food Frequency Questionnaire to assess for changes over the 1 year follow up period.
Cross-over and contamination in the control arm - Physical Activity levels | 1 Year
  Changes in physical activity will be monitored using the International Physical Activity Questionnaire, which is used to calculate total metabolic equivalent task (MET) minutes.
Cross-over and contamination in the control arm - Psychological Health Activities | 1 Year
  Measured by the number of participants in the control arm who perform activities in which the goal of the activity was to improve mental and emotional health.

SECONDARY OUTCOMES:
Communication | 2 years
  Assessing the type and frequency of communications between research staff at The Ottawa Hospital (TOH) and the Centre for Health Innovation (CHI), as well as within TOH and the CHI through number of emails, phone calls, meetings (in-person or virtual) or any other communication method.
Natural Killer Cell Function | Enrolment, 2-3 days pre-op, and 6 months and 12 months post surgery
  Measured by serum Interferon Gamma Levels
Qualitative Experience | 2 years
  Evaluate the qualitative experience of care of participants in both arms through semi-structured interviews
Inflammatory Response | Enrolment, 2-3 days pre-op, and 1 day, 3-4 weeks, 6 months, and 12 months post-surgery
  Measured by serum C-Reactive Protein Levels
Neutrophil to Lymphocyte Ratio | Enrolment, 2-3 days pre-op, and 6 months and 12 months post surgery
  Measured by collecting a complete blood count with differential and comparing neutrophil and lymphocyte levels

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Seely, MD, PhD, FRCSC, Principal Investigator — Ottawa Hospital Research Institute; Dugald Seely, ND, MSc, Principal Investigator — The Canadian College of Naturopathic Medicine
Locations (2):
- Canada (2):
  - The Ottawa Hospital, Ottawa, Ontario
  - Michael Garron Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No